CLINICAL TRIAL: NCT03391479
Title: A Phase 2, Multi-centre, Open-label Study of Avelumab (MSB0010718C) in Locally Advanced or Metastatic Penile Cancer Patients Unfit for Platinum-based Chemotherapy or Progressed On or After Platinum-based Chemotherapy
Brief Title: A Study of Avelumab in Penile Cancer Who Are Unfit for or Have Progressed After Platinum-Based Chemotherapy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALPACA; 17-6013 (Other: UHN)
Record Dates: First submitted 2017-12-29; First posted 2018-01-05 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Penile Cancer; Advanced Cancer; Metastatic Cancer
MeSH Terms: conditions — Penile Neoplasms; Neoplasm Metastasis | interventions — avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Avelumab and Best Supportive Care (Experimental): Avelumab will be given intravenously (by vein) at a dose of 10 mg/kg, once every 2 weeks
  Best supportive care will be provided as required.
  Interventions: Drug: Avelumab; Other: Best Supportive Care

INTERVENTIONS:
Drug: Avelumab — Avelumab is a fully human monoclonal antibody (mAb) of the immunoglobulin (Ig) G1 isotype. Avelumab selectively binds to programmed death-ligand 1 (PD-L1) and competitively blocks its interaction with programmed death protein 1 (PD-1).
Other: Best Supportive Care — As required.

SUMMARY:
This is a phase 2 study whose purpose is see how useful investigational drug, avelumab, is in patients with locally advanced or metastatic penile cancer who are unfit for or progressed on platinum-based chemotherapy.

The usefulness of avelumab in this study population will be determined by anti-tumor activity assessed by objective response rate.

Avelumab is a monoclonal antibody that binds to a protein called programmed death-ligand 1 (PD-L1) and blocks its communication with another protein called programmed death protein 1 (PD-1). The communication of these proteins are thought to be important in the growth of tumors. Blocking these proteins from communicating may stop or shrink tumors.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed squamous cell carcinoma of the penis
* Measurable disease per Immune-related Response Evaluation Criteria in Solid Tumors (iRECIST)
* Unresectable/metastatic disease that is unfit for platinum-based chemotherapy OR disease that has progressed on or after treatment with platinum-based chemotherapy
* ≥18 years of age
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2

Exclusion Criteria:

* Prior immunotherapy with IL-2, IFN-α, or an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or CTLA-4 antibody (including ipilimumab), or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways
* Major surgery ≤4 weeks or major radiation therapy ≤2 weeks prior to enrollment
* Known symptomatic central nervous system (CNS) metastases requiring steroids
* Active autoimmune disease that might deteriorate when receiving an immunostimulatory agent
* Diagnosis of prior immunodeficiency or organ transplant requiring immunosuppressive therapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 25 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | 4 weeks
  To demonstrate the anti-tumor activity of avelumab by objective response rate (ORR) according to Immune-related Response Evaluation Criteria in Solid Tumors (iRECIST) in patients with locally advanced or metastatic penile carcinoma unfit for platinum-based chemotherapy or progressed on or after platinum-based chemotherapy.

SECONDARY OUTCOMES:
Progression-free Survival Rate | 3 years
  Assess the progression free survival (PFS) of avelumab in patients determined to have PD-L1-positive tumors (including infiltrating immune cells) by the GMP verified Dako PD-L1 IHC 22C3 pharmDx test with thresholds of <1%, 1-49%, and ≥ 50% to define PD-L1 positivity, and in all enrolled patients
Overall Survival Rate | 3 years
  Assess the overall survival (OS) of avelumab in patients determined to have PD-L1-positive tumors (including infiltrating immune cells) by the GMP verified Dako PD-L1 IHC 22C3 pharmDx test with thresholds of <1%, 1-49%, and ≥ 50% to define PD-L1 positivity, and in all enrolled patients

CONTACTS AND LOCATIONS:
Overall Officials: Srikala Sridhar, M.D., Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada